CLINICAL TRIAL: NCT03895593
Title: Rescue Fecal Microbiota Transplantation for Refractory Intestinal Infections: China National Registry
Brief Title: Rescue Fecal Microbiota Transplantation for National Refractory Intestinal Infections
Status: Recruiting | Type: Observational
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Second Affiliated Hospital of Suzhou University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Shenzhen Hospital of Southern Medical University (Other); Wuhan University (Other); LiuZhou People's Hospital (Other); Lishui Country People's Hospital (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, The Second Hospital of Nanjing Medical University
Other Study IDs: FMT-CN-190321
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2019-03

CONDITIONS: Intestinal Infection; Clostridioides Difficile Infection; Antibiotic-associated Diarrhea
Keywords: fecal microbiota transplantation; intestinal infection; clostridioides Difficile Infection; Antibiotic-associated Diarrhea; Washed microbiota transplantation
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: rescue fecal microbiota transplantation — Fecal microbiota transplantation refers to the infusion of fecal microbiota from healthy donor into patients' gastrointestinal tract. The delivering ways for FMT include but are not limited to gastroscopy, colonoscopy, edema, nasogastric tube, transendoscopic enteral tube, and etc.

SUMMARY:
A national data registry of patients receiving the rescue fecal microbiota transplantation for the refractory intestinal infections from the China Microbiota Transplantation System was designed to assess the short-term and long-term safety and efficacy.

DETAILED DESCRIPTION:
This registry will enroll national patients with refractory intestinal infections (including clostridioides difficile infection, other infections with known or unknown pathogens) receiving rescue fecal microbiota transplantation (FMT) from the the China Microbiota Transplantation System. The improved methodology of FMT based on the automatic washing process and the related delivering consideration was named as washed microbiota transplantation (WMT) by the consensus statement from the FMT-standardization study group in 2019.12. Data of demographic characteristics, symptoms of intestinal infections, previous medicine treatment and clinical outcomes will be collected retrospectively abstracted from the electronic medical records or prospective follow-up. All the patients will be followed up for at least 12 weeks post-FMT. Information on follow-up will be designed to assess the short-term and long-term adverse events.

ELIGIBILITY:
Inclusion Criteria: National patients with refractory intestinal infections receiving rescue FMT from the China Microbiota Transplantation System from September 2015 to December, 2029 will be included.

-

Exclusion Criteria: Patients will be excluded from the analysis if they are not followed up for at least 12 weeks post-FMT.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: National patients with refractory intestinal infections receiving rescue FMT from the Chinese fmtBank from September, 2015 to December, 2029 will be included
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09-25 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
abdominal symptom outcomes | 1 week
  Definitions used to classify response, nonresponse and exacerbation for the abdominal symptom outcomes are based on the physicians' holistic evaluation of patients' abdominal symptoms.
survival outcome | 4 weeks
  The survival outcome refers to the 4-week survival post-FMT.
clinical cure of clostridioides difficile infection | 8 weeks
  clinical resolution (absence of diarrhea, or marked reduction in stool frequency), or a negative clostridioides difficile (CD) test, without the need for further anti-clostridioides difficile infection therapy

SECONDARY OUTCOMES:
adverse events | 12 weeks
  Unfavorable signs, symptoms, or major changes from pre-FMT laboratory test results.

CONTACTS AND LOCATIONS:
Overall Officials: faming zhang, MD,PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang F, Cui B, He X, Nie Y, Wu K, Fan D; FMT-standardization Study Group. Microbiota transplantation: concept, methodology and strategy for its modernization. Protein Cell. 2018 May;9(5):462-473. doi: 10.1007/s13238-018-0541-8. Epub 2018 Apr 24. PMID 29691757
- [Background] McDonald D, Ackermann G, Khailova L, Baird C, Heyland D, Kozar R, Lemieux M, Derenski K, King J, Vis-Kampen C, Knight R, Wischmeyer PE. Extreme Dysbiosis of the Microbiome in Critical Illness. mSphere. 2016 Aug 31;1(4):e00199-16. doi: 10.1128/mSphere.00199-16. eCollection 2016 Jul-Aug. PMID 27602409
- [Background] Li Q, Wang C, Tang C, He Q, Zhao X, Li N, Li J. Successful treatment of severe sepsis and diarrhea after vagotomy utilizing fecal microbiota transplantation: a case report. Crit Care. 2015 Feb 9;19(1):37. doi: 10.1186/s13054-015-0738-7. PMID 25881250
- [Background] Litao G, Jingjing S, Yu L, Lei Z, Xiaona H, Zhijing Z. Risk Factors for Antibiotic-Associated Diarrhea in Critically Ill Patients. Med Sci Monit. 2018 Jul 18;24:5000-5007. doi: 10.12659/MSM.911308. PMID 30020891
- [Background] van Beurden YH, Nieuwdorp M, van de Berg PJEJ, Mulder CJJ, Goorhuis A. Current challenges in the treatment of severe Clostridium difficile infection: early treatment potential of fecal microbiota transplantation. Therap Adv Gastroenterol. 2017 Apr;10(4):373-381. doi: 10.1177/1756283X17690480. Epub 2017 Feb 8. PMID 28491142
- [Background] Wei Y, Yang J, Wang J, Yang Y, Huang J, Gong H, Cui H, Chen D. Successful treatment with fecal microbiota transplantation in patients with multiple organ dysfunction syndrome and diarrhea following severe sepsis. Crit Care. 2016 Oct 18;20(1):332. doi: 10.1186/s13054-016-1491-2. PMID 27751177
- [Derived] Wu X, Ai RJ, Xu J, Wen Q, Pan HQ, Zhang ZH, Ning W, Fang Y, Ding DF, Wang Q, Han S, Liu X, Wu M, Jia ZY, Jia S, Lin T, Cui BT, Nie YZ, Wang X, Zhang FM. Washed microbiota transplantation for Clostridioides difficile infection: A national multicenter real-world study. J Dig Dis. 2023 Oct;24(10):540-549. doi: 10.1111/1751-2980.13227. Epub 2023 Oct 5. PMID 37681235
- [Derived] Dai M, Liu Y, Chen W, Buch H, Shan Y, Chang L, Bai Y, Shen C, Zhang X, Huo Y, Huang D, Yang Z, Hu Z, He X, Pan J, Hu L, Pan X, Wu X, Deng B, Li Z, Cui B, Zhang F. Rescue fecal microbiota transplantation for antibiotic-associated diarrhea in critically ill patients. Crit Care. 2019 Oct 21;23(1):324. doi: 10.1186/s13054-019-2604-5. PMID 31639033